CLINICAL TRIAL: NCT05797415
Title: Sentinel Lymph Node Biopsy in Ocular Surface and Adnexal Cancers: Prospective Observational Study
Brief Title: Sentinel Lymph Node Biopsy in Ocular Surface and Adnexal Cancers
Acronym: BLS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Savino Gustavo, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5572
Record Dates: First submitted 2023-03-06; First posted 2023-04-04 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ocular Sebaceous Carcinoma; Ocular Basal Cell Carcinoma; Ocular Surface Squamous Neoplasia; Merkel Cell Carcinoma, Unspecified; Porocarcinoma; Conjunctival Melanoma
Keywords: Sentinel Lymph Node Biopsy; Malignant ocular surface tumors; Malignant eyelids tumors
MeSH Terms: conditions — Carcinoma, Merkel Cell; Eccrine Porocarcinoma | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Sebaceous carcinoma: patients with sebaceous carcinoma both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A. Gemelli IRCCS
  Interventions: Procedure: Sentinel Lymph Node Biopsy
- Merkel's carcinoma: patients with Merkel's carcinoma both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A. Gemelli IRCCS
  Interventions: Procedure: Sentinel Lymph Node Biopsy
- Porocarcinoma: patients with Porocarcinoma both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A. Gemelli IRCCS
  Interventions: Procedure: Sentinel Lymph Node Biopsy
- Conjunctival Melanoma: patients with Conjunctival Melanoma both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A. Gemelli IRCCS
  Interventions: Procedure: Sentinel Lymph Node Biopsy
- Squamous cell Carcinoma: patients with squamous cell Carcinoma of the ocular surface and adnexa both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A. Gemelli IRCCS
  Interventions: Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — * Injection of 99mTc-labeled nanocolloids
  * Preoperative lymphoscintigraphy
  * Intraoperative gamma probe search of the sentinel lymph node
  * Sentinel lymph node biopsy
  * Excisional biopsy of the neoformation in cases not undergoing excision before SLN biopsy.
  * If the SLN is histologically positive, the multidisciplinary team will consider whether to refer the patient for parotidectomy and excision of the lymph node chain and/or adjuvant radio/chemotherapy.

SUMMARY:
The study involves enrollment of patients with sebaceous carcinoma, Merkel's carcinoma, Porocarcinoma, Melanoma, and squamous cell Ca of the ocular surface and adnexa both primary and relapsed after surgical and/or radiation-chemotherapy treatment at the Fondazione Policlinico Universitario A. Gemelli, IRCCS. The study will last 9 years: 1 year will be devoted to the first phase of the study. Patient enrollment will continue for an additional 3 years, and 5 years will be devoted overall to patient follow-up so that survival outcomes at 1-3 and 5 years can be assessed in a congruent number of patients. A preliminary analysis of the data at 1 year (pilot phase), an analysis at 4 years to confirm the preliminary study data on a larger sample, and a final analysis to evaluate OS and PFS at the 3 time-points indicated are planned.

DETAILED DESCRIPTION:
Patients will undergo:

* Evaluation in the ocular oncology outpatient clinic with examination and anterior segment photography
* Staging according to TNM AJCC 8th edition by incisional biopsy (if necessary after clinical evaluation) and/or excisional biopsy and imaging to be performed in current clinical practice (MRI with mdc orbits, massif and neck + Tc/Pet total body)
* Injection of 99mTc-labeled nanocolloids
* Preoperative lymphoscintigraphy
* Intraoperative search by gamma probe of the sentinel lymph node
* Sentinel lymph node biopsy
* Excisional biopsy of the neoformation in cases not undergoing excision before SLN biopsy.
* In case of SLN histologic positivity, the multidisciplinary team will consider whether to refer the patient for parotidectomy and excision of the lymph node chain and/or adjuvant radio/chemotherapy.
* Clinical-instrumental follow-up to be performed in current clinical practice (Clinical examination, cranial orbit and neck MRI, total body CT scan) at 3, 6, 12, 18, 24, 36, 48, 60 months or according to periodicity assessed on a case-by-case basis by the Tumor Board.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Porocarcinoma, Ca of Merkel, Ca Sebaceous
* Patients with cutaneous adnexal melanoma with thickness ≥1.5 mm, Clark's level ≥3, >1 mitotic figure per high-power field.
* Patients with conjunctival melanoma both primary and recurrent and associated with primary acquired melanosis with atypia.
* Patients with squamous cell Ca of adnexa with Staging ≥3, locally recurrent or with perineural invasion
* Patients with squamous cell Ca of the surface with Staging ≥3 and/or multicenter
* Signature of informed consent to participate in the study
* cNo

Exclusion Criteria:

* Age less than 18 years
* Patients with metastatic disease at diagnosis
* All patients who do not fit the inclusion criteria
* Failure to obtain informed consent

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with sebaceous carcinoma, Merkel's carcinoma, Porocarcinoma, Melanoma, and squamous cell Ca of the ocular surface and adnexa both primary and relapsed after surgical and/or radiation-chemotherapy treatment at Fondazione Policlinico Universitario A.Gemelli IRCCS will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2032-03-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of lymphoscintigraphic examination and SLN biopsy | 9 years
  Positive predictive value (PPV) and negative predictive value (NPV), in percentage, in order to determine the likelihood of lymphoscintigraphic examination and SLN biopsy in diagnosing Ocular Surface and Adnexal Cancers.
Efficacy of lymphoscintigraphic examination and SLN biopsy | 9 years
  Sensitivity and sensibility, in percentage, in order to determine the likelihood of lymphoscintigraphic examination and SLN biopsy in diagnosing Ocular Surface and Adnexal Cancers.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  OS (in years) at 1, 3, and 5 years
Diseases Free Survival (DFS) | 5 years
  DFS (in years) at 1,3 and 5 years
Progression Free Survival (PFS) | 5 years
  PFS (in years) at 1, 3, and 5 years
Changes in clinical parameter (tumor diameters) | 60 months
  Changes in clinical parameter (tumor diameters) of patients at follow-up (3, 6, 12, 24, 36, 48, 60 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavo Savino, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields CL, Alset AE, Boal NS, Casey MG, Knapp AN, Sugarman JA, Schoen MA, Gordon PS, Douglass AM, Sioufi K, Say EA, Shields JA. Conjunctival Tumors in 5002 Cases. Comparative Analysis of Benign Versus Malignant Counterparts. The 2016 James D. Allen Lecture. Am J Ophthalmol. 2017 Jan;173:106-133. doi: 10.1016/j.ajo.2016.09.034. Epub 2016 Oct 8. PMID 27725148
- [Background] Shields CL, Shields JA. Tumors of the conjunctiva and cornea. Indian J Ophthalmol. 2019 Dec;67(12):1930-1948. doi: 10.4103/ijo.IJO_2040_19. PMID 31755426
- [Background] Esmaeli B, Wang B, Deavers M, Gillenwater A, Goepfert H, Diaz E, Eicher S. Prognostic factors for survival in malignant melanoma of the eyelid skin. Ophthalmic Plast Reconstr Surg. 2000 Jul;16(4):250-7. doi: 10.1097/00002341-200007000-00002. PMID 10923972
- [Background] Soysal HG, Markoc F. Invasive squamous cell carcinoma of the eyelids and periorbital region. Br J Ophthalmol. 2007 Mar;91(3):325-9. doi: 10.1136/bjo.2006.102673. Epub 2006 Oct 4. PMID 17020898
- [Background] Faustina M, Diba R, Ahmadi MA, Esmaeli B. Patterns of regional and distant metastasis in patients with eyelid and periocular squamous cell carcinoma. Ophthalmology. 2004 Oct;111(10):1930-2. doi: 10.1016/j.ophtha.2004.02.009. PMID 15465559
- [Background] Cervantes G, Rodriguez AA Jr, Leal AG. Squamous cell carcinoma of the conjunctiva: clinicopathological features in 287 cases. Can J Ophthalmol. 2002 Feb;37(1):14-9; discussion 19-20. doi: 10.1016/s0008-4182(02)80093-x. PMID 11865953
- [Background] Yousef YA, Finger PT. Squamous carcinoma and dysplasia of the conjunctiva and cornea: an analysis of 101 cases. Ophthalmology. 2012 Feb;119(2):233-40. doi: 10.1016/j.ophtha.2011.08.005. Epub 2011 Dec 20. PMID 22189448
- [Background] Esmaeli B, Eicher S, Popp J, Delpassand E, Prieto VG, Gershenwald JE. Sentinel lymph node biopsy for conjunctival melanoma. Ophthalmic Plast Reconstr Surg. 2001 Nov;17(6):436-42. doi: 10.1097/00002341-200111000-00010. PMID 11766025
- [Background] Freitag SK, Aakalu VK, Tao JP, Wladis EJ, Foster JA, Sobel RK, Yen MT. Sentinel Lymph Node Biopsy for Eyelid and Conjunctival Malignancy: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 Dec;127(12):1757-1765. doi: 10.1016/j.ophtha.2020.07.031. Epub 2020 Jul 19. PMID 32698034
- [Background] Chak G, Morgan PV, Joseph JM, Tao JP. A positive sentinel lymph node in periocular invasive squamous cell carcinoma: a case series. Ophthalmic Plast Reconstr Surg. 2013 Jan-Feb;29(1):6-10. doi: 10.1097/IOP.0b013e31826a50f7. PMID 23034693
- [Background] Maalouf TJ, Dolivet G, Angioi KS, Leroux A, Genin P, George JL. Sentinel lymph node biopsy in patients with conjunctival and eyelid cancers: experience in 17 patients. Ophthalmic Plast Reconstr Surg. 2012 Jan-Feb;28(1):30-4. doi: 10.1097/IOP.0b013e31822fb44b. PMID 22262287
- [Background] Savino G, Cuffaro G, Maceroni M, Pagliara MM, Sammarco MG, Giraldi L, Blasi MA. Advanced ocular surface squamous cell carcinoma (OSSC): long-term follow-up. Graefes Arch Clin Exp Ophthalmol. 2021 Nov;259(11):3437-3443. doi: 10.1007/s00417-021-05264-3. Epub 2021 Jul 20. PMID 34283293
- [Background] Esmaeli B, Nasser QJ, Cruz H, Fellman M, Warneke CL, Ivan D. American Joint Committee on Cancer T category for eyelid sebaceous carcinoma correlates with nodal metastasis and survival. Ophthalmology. 2012 May;119(5):1078-82. doi: 10.1016/j.ophtha.2011.11.006. Epub 2012 Feb 11. PMID 22330966